CLINICAL TRIAL: NCT00861224
Title: The Effects of Long-term Dosing of AMG 531 on Bone Marrow Morphology in Thrombocytopenic Subjects With Immune (Idiopathic) Thrombocytopenic Purpura (ITP)
Brief Title: Effects of Long-term Dosing of AMG 531 on Bone Marrow Morphology
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Other Study IDs: 20050123
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biospecimen samples were retained.

GROUPS / COHORTS (1):
- Observed Subjects: Subjects that submitted bone marrow biopsy and aspirates.
  Interventions: Other: No Intervention for Observational Study

INTERVENTIONS:
Other: No Intervention for Observational Study — No intervention was used on this protocol, as this was an observational study.

SUMMARY:
This study was conducted in conjunction with the 2 phase 3 studies of AMG 531 (20030105 and 20030212) and an open-label extension study (20030213) and compared pretreatment and posttreatment bone marrow samples for the purpose of studying morphologic changes.

DETAILED DESCRIPTION:
This study is to be performed in conjunction with the phase 3 treatment studies (20030105 and 20030212) and with the open label extension study (20030213).

Subjects who are screening for participation in the phase 3 studies will be asked to consider participation in this bone marrow study. At least 10 subjects from each of the two phase 3 studies (20030105 and 20030212) will enroll in this study. This will ensure enrollment of subjects who are both non-splenectomized and splenectomized.

All subjects who participate must have had a bone marrow biopsy within one year prior to enrollment, and must release the tissue block to Amgen for interpretation by a central pathology laboratory. Subjects that do not have a historical bone marrow within one year (with available tissue block) must have a baseline bone marrow biopsy and aspirate performed prior to dosing with AMG 531.

Subjects will be assigned to a follow-up bone marrow biopsy and aspirate after either 9 months or 6 months of treatment. The subjects will be assigned to follow-up time in descending order, with the first 5 subjects from each study assigned to 9 month follow-up, and the last 5 subjects from each study assigned to 6 month follow-up. Some subjects will have their follow-up bone marrow biopsy and aspirate while on the open label extension study (20030213).

To eliminate the possibility of performing a bone marrow biopsy and aspirate on a placebo subject, all subjects who were assigned to a 6 month follow-up will be unblinded at the end of the phase 3 study treatment period (week 26). If the subject was on AMG 531, they must have their follow-up bone marrow biopsy and aspirate within one week (week 27). If the subject was on placebo, they will have their follow-up bone marrow performed after 3 months of treatment in the open label study.

The subjects that were assigned to a 9 month follow-up will have their platelet counts monitored as required by the phase 3 protocol. Any subject who has a platelet count > 50 x 109/L at week 26 of the phase 3 study, will be required to schedule a bone marrow biopsy and aspirate for week 27. If their platelet count is still > 50 x 109/L at week 27, they will have their bone marrow biopsy and aspirate at that time. If their platelet count drops to ≤ 50 x 109/L prior to week 27, they will have their follow-up bone marrow biopsy and aspirate performed after completing 3 months of treatment on the open label study (20030213).

Subjects who discontinue AMG 531 treatment will have the follow-up bone marrow biopsy and aspirate at the time of discontinuation, regardless of the pre-assigned date of the follow-up.

If a subject requires a bone marrow biopsy and aspirate as part of a safety assessment, this assessment will be counted as the follow-up bone marrow biopsy regardless of the timing of the assessment. Any additional clinically warranted bone marrow biopsies will also be sent to the central pathology lab for review.

All bone marrow biopsy reports will be provided by the central lab at the end of this study, but will not be available for clinical management at the time that the sample is collected.

All bone marrow biopsies will be evaluated by the central pathology lab.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be enrolled in AMG 531 protocol 20030105 or 20030212
* Subject must have had a bone marrow biopsy within one year of enrollment (with available tissue block to send to a central pathology laboratory for interpretation) or must consent to a pre-treatment bone marrow biopsy and aspirate
* Written informed consent

Exclusion Criteria:

* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Splenectomized or nonsplenectomized subjects with a primary diagnosis of ITP from either of the phase 3 studies (20030105 or 20030212) or the open-label extension study 20030213; pretreatment bone marrow biopsy within 1 year of enrollment into the phase 3 study; separate written informed consent for the follow-up bone marrow.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2005-08; Primary Completion 2006-10 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The changes from baseline in bone marrow morphology by subject | Entire duration of the study

SECONDARY OUTCOMES:
The changes from baseline in bone marrow morphology by dose range | Entire duration of the study
The changes from baseline in bone marrow morphology by length of treatment with AMG 531 | Entire duration of the study
The changes from baseline bone marrow morphology for splenectomized and non-splenectomized subjects | Entire duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Kuter DJ, Mufti GJ, Bain BJ, Hasserjian RP, Davis W, Rutstein M. Evaluation of bone marrow reticulin formation in chronic immune thrombocytopenia patients treated with romiplostim. Blood. 2009 Oct 29;114(18):3748-56. doi: 10.1182/blood-2009-05-224766. Epub 2009 Aug 11. PMID 19671919
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_46_AMP-2_20050123.pdf
- See also: FDA-approved Drug Labeling — http://www.nplate.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com